CLINICAL TRIAL: NCT04709835
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Antiviral Activity, Safety, Pharmacokinetics, and Efficacy of RO7496998 (AT-527) in Non-Hospitalized Adult Patients With Mild or Moderate COVID-19
Brief Title: Study to Evaluate the Effects of AT-527 in Non-Hospitalized Adult Patients With Mild or Moderate COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WV43042; 2020-005366-34 (EudraCT Number)
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Results first posted 2022-10-13 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — AT-511

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive AT-527-matched placebo twice a day (BID) on Days 1-5.
  Interventions: Drug: Placebo
- AT-527 550 mg (1x550 mg) (Experimental): Participants will receive 550 mg AT-527 (1x550 mg) twice a day (BID) on Days 1-5.
  Interventions: Drug: AT-527
- AT-527 1100 mg (4x275 mg) (Experimental): Participants will receive 1100 mg AT-527 (4x275 mg) twice a day (BID) on Days 1-5.
  Interventions: Drug: AT-527

INTERVENTIONS:
Drug: AT-527 — Results from Arm AT-527 500 mg determined the dose and regimen to be used for AT-527 1100 mg.
  Other Names: RO7496998
  Arms: AT-527 1100 mg (4x275 mg); AT-527 550 mg (1x550 mg)
Drug: Placebo — The dose and regimen of the placebo will match that of the respective AT-527 comparator arm.
  Arms: Placebo

SUMMARY:
This randomized study evaluates the antiviral activity, safety, efficacy and pharmacokinetics of AT-527 versus a placebo in participants with mild or moderate coronavirus disease (COVID-19) who are not hospitalized.

ELIGIBILITY:
Inclusion Criteria:

* Positive SARS-CoV-2 diagnostic test (RT-PCR or rapid antigen test)at screening
* Has symptoms consistent with mild or moderate COVID-19, as determined by the investigator, with onset ≤5 days prior to randomization

Exclusion Criteria:

* Clinical signs indicative of COVID-19 illness requiring hospitalization, defined as any of the following: shortness of breath at rest, respiratory rate ≥30, heart rate ≥125, peripheral capillary oxygen saturation ≤93% on room air
* Treatment with a therapeutic agent against SARS-CoV-2 including, but not limited to, other direct acting antivirals, convalescent plasma, monoclonal antibodies against SARS CoV-2, or intravenous immunoglobulin within 3 months or less than 5 drug elimination half-lives (whichever is longer) prior to screening
* Requirement, in the opinion of the investigator, for any of the prohibited medications during the study
* Use of hydroxychloroquine or amiodarone within 3 months of screening
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 30 days after the final dose of AT-527. Women of childbearing potential must have a negative urine pregnancy test result at screening
* Abnormal laboratory test results at screening
* Clinically significant abnormal ECG, as determined by the Investigator, at screening
* Planned procedure or surgery during the study
* Known allergy or hypersensitivity to study drug or drug product excipients
* Substance abuse, as determined by the investigator, within 12 months prior to screening
* Poor peripheral venous access
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* Any clinically significant history of epistaxis within the last 3 months and/or history of being hospitalized due to epistaxis of any previous occasion
* History of anaphylaxis
* Any uncontrolled serious medical condition or other clinically significant abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- Hamilton Medical Research Group, Hamilton, Ontario, Canada
- Greece (2):
  - National and Kapodistrian University of Athens, Athens
  - General State Hospital of Nikaia St Panteleimon, Nikaia Attikis
- Connolly Hospital, Dublin, Ireland
- Latvia (2):
  - Outpatient Clinic Adoria, Riga
  - The Family Physician's Practice of Dr. Maija Kozlovska, Salaspils
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
- United Kingdom (4):
  - Chapel Street Medical Centre, Ashton-under-Lyne
  - Tower Family Healthcare - Moorgate Primary Care Ce, Bury
  - CPS Research, Glasgow
  - Chelsea and Westminster NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm)

REFERENCES:
- [Derived] Boffito M, Dolan E, Singh K, Holmes W, Wildum S, Horga A, Pietropaolo K, Zhou XJ, Clinch B, Collinson N, Ukachukwu V. A Phase 2 Randomized Trial Evaluating the Antiviral Activity and Safety of the Direct-Acting Antiviral Bemnifosbuvir in Ambulatory Patients with Mild or Moderate COVID-19 (MOONSONG Study). Microbiol Spectr. 2023 Aug 17;11(4):e0007723. doi: 10.1128/spectrum.00077-23. Epub 2023 Jun 20. PMID 37338393

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at sites in the United Kingdom, Spain, Greece, Latvia, Ireland and Canada.
Pre-assignment Details: The study enrolled non-hospitalized adult participants with mild or moderate COVID-19. Four enrolled participants were not treated and are not included in the Results.
Groups:
- Pooled Placebo: Participants received placebo matched to 550 mg or 1100 mg AT-527 twice a day (BID) on Days 1-5.
- AT-527 550 mg (1x550 mg): Participants received 550 mg AT-527 (1x550 mg) twice a day (BID) on Days 1-5.
- AT-527 1100 mg (4x275 mg): Participants received 1100 mg AT-527 (4x275 mg) twice a day (BID) on Days 1-5.
Period: Overall Study
Arm/Group | Pooled Placebo | AT-527 550 mg (1x550 mg) | AT-527 1100 mg (4x275 mg)
Started | 40 | 30 | 30
Completed | 40 | 29 | 30
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The modified ITT infected (mITTi) population was defined as all participants randomized in the study who received any amount of study drug and had at least one positive SARS-CoV-2 RT-PCR test result above or equal to the limit of quantification (LOQ) during the study, with participants grouped according to the treatment assignment at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | AT-527 550 mg (1x550 mg) | AT-527 1100 mg (4x275 mg) | Total
Number analyzed (Participants) | 40 | 30 | 30 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (13.2) | 32.7 (10.9) | 40.3 (15.6) | 36.6 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 15 | 17 | 54
  Male | 18 | 15 | 13 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 1 | 8
  Not Hispanic or Latino | 36 | 26 | 29 | 91
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 3
  White | 38 | 29 | 28 | 95
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Amount of Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Virus RNA at Baseline [Mean (Standard Deviation); unit: log10 copies/mL] — SARS-CoV-2 virus RNA was measured by reverse-transcription polymerase chain reaction (RT-PCR).
  log10 copies/mL | 6.24 (1.40) | 6.98 (1.10) | 5.94 (1.46) | 6.37 (1.39)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Amount of Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Virus RNA for AT-527 550 mg and Matched Placebo
Description: SARS-CoV-2 virus RNA was measured by reverse-transcription polymerase chain reaction (RT-PCR) from nasopharyngeal (NP) swabs. The change from baseline was estimated from an ANCOVA model with baseline viral load as a covariate. Reported here is the adjusted mean change from baseline. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Day 3, Day 5, Day 7
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: log10 copies/mL
Groups:
- Placebo Matched to AT-527 550 mg: Participants received placebo matched to 550 mg AT-527 twice a day (BID) on Days 1-5.
Arm/Group | Placebo Matched to AT-527 550 mg | AT-527 550 mg (1x550 mg)
Number analyzed (Participants) | 30 | 30
log10 copies/mL
  Day 3: number analyzed (Participants) | 30 | 29
  Day 3 | -1.16 (0.203) | -1.26 (0.206)
  Day 5: number analyzed (Participants) | 29 | 30
  Day 5 | -2.42 (0.230) | -2.11 (0.226)
  Day 7: number analyzed (Participants) | 29 | 29
  Day 7 | -3.13 (0.220) | -3.38 (0.220)
Statistical Analysis 1: Comparison: Placebo Matched to AT-527 550 mg vs AT-527 550 mg (1x550 mg); Day 3; Test type: Superiority; p = 0.7144, ANCOVA; Difference in Adjusted Means = -0.11, 80% CI 2-sided [-0.49 to 0.27], Standard Error of Mean 0.292 — A difference in adjusted means of <0 favors RO7496998 (AT-527)
Statistical Analysis 2: Comparison: Placebo Matched to AT-527 550 mg vs AT-527 550 mg (1x550 mg); Day 5; Test type: Superiority; p = 0.3373, ANCOVA; Difference in Adjusted Means = 0.32, 80% CI 2-sided [-0.11 to 0.74], Standard Error of Mean 0.327 — A difference in adjusted means of <0 favors RO7496998 (AT-527)
Statistical Analysis 3: Comparison: Placebo Matched to AT-527 550 mg vs AT-527 550 mg (1x550 mg); Day 7; Test type: Superiority; p = 0.4260, ANCOVA; Difference in Adjusted Means = -0.25, 80% CI 2-sided [-0.66 to 0.16], Standard Error of Mean 0.315 — A difference in adjusted means of <0 favors RO7496998 (AT-527)

2. Secondary Outcome: Time to Cessation of SARS-CoV-2 Viral Shedding
Description: Time to cessation of viral shedding was defined as the time between the initiation of any study treatment and the first time when a negative or below the limit of detection RT-PCR test result was obtained. RT-PCR was measured from NP swabs. Median, 25th and 75th percentiles were estimated from the Kaplan-Meier curve.
Time Frame: Up to Day 7
Population: The mITTi population was defined as all participants randomized in the study who received any amount of study drug and had at least one positive SARS-CoV-2 RT-PCR test result above or equal to the limit of quantification (LOQ) during the study, with participants grouped according to the treatment assignment at randomization.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Pooled Placebo | AT-527 550 mg (1x550 mg) | AT-527 1100 mg (4x275 mg)
Number analyzed (Participants) | 40 | 30 | 30
hours | NA [144.2 to NA] — NA = Not estimable due to low number of participants with event. | NA [143.8 to NA] — NA = Not estimable due to low number of participants with event. | NA [141.1 to NA] — NA = Not estimable due to low number of participants with event.
Statistical Analysis 1: Comparison: Pooled Placebo vs AT-527 550 mg (1x550 mg); Test type: Superiority; Hazard Ratio (HR) = 0.96, 80% CI 2-sided [0.53 to 1.74] — Hazard ratio (80% CI) was estimated with a Cox proportional hazards model (unadjusted)
Statistical Analysis 2: Comparison: Pooled Placebo vs AT-527 1100 mg (4x275 mg); Test type: Superiority; Hazard Ratio (HR) = 1.33, 80% CI 2-sided [0.76 to 2.32] — Hazard ratio (80% CI) was estimated with a Cox proportional hazards model (unadjusted)

3. Secondary Outcome: Time to Sustained Non-Detectable SARS-CoV-2 Virus RNA
Description: Time to sustained non-detectable SARS-CoV-2 virus RNA was defined as the time between the initiation of any study treatment and first time when a negative or below the limit of detection test result by RT-PCR is obtained after which no positive test above or equal to the limit of detection was reported. RT-PCR was measured from NP swabs. Median, 25th and 75th percentiles were estimated from the Kaplan-Meier curve.
Time Frame: Up to Day 7
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Pooled Placebo | AT-527 550 mg (1x550 mg) | AT-527 1100 mg (4x275 mg)
Number analyzed (Participants) | 40 | 30 | 30
hours | NA [NA to NA] — NA = Not estimable due to low number of participants with event. | NA [NA to NA] — NA = Not estimable due to low number of participants with event. | NA [NA to NA] — NA = Not estimable due to low number of participants with event.
Statistical Analysis 1: Comparison: Pooled Placebo vs AT-527 550 mg (1x550 mg); Test type: Superiority; Hazard Ratio (HR) = 0.86, 80% CI 2-sided [0.44 to 1.70] — Hazard ratio (80% CI) was estimated with a Cox proportional hazards model (unadjusted)
Statistical Analysis 2: Comparison: Pooled Placebo vs AT-527 1100 mg (4x275 mg); Test type: Superiority; Hazard Ratio (HR) = 1.06, 80% CI 2-sided [0.56 to 2.03] — Hazard ratio (80% CI) was estimated with a Cox proportional hazards model (unadjusted)

4. Secondary Outcome: Percentage of Participants Positive for SARS-CoV-2 Virus RNA at Specified Timepoints
Description: Reported here is the percentage of participants with a positive virus RNA by RT-PCR test result above or equal to the limit of quantification (LOQ). RT-PCR was measured from NP swabs.
Time Frame: Baseline, Day 3, Day 5, Day 7
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo | AT-527 550 mg (1x550 mg) | AT-527 1100 mg (4x275 mg)
Number analyzed (Participants) | 40 | 30 | 30
percentage of participants
  Baseline | 100 | 100 | 96.7
  Day 3: number analyzed (Participants) | 40 | 30 | 29
  Day 3 | 95.0 | 100 | 93.1
  Day 5: number analyzed (Participants) | 38 | 30 | 30
  Day 5 | 84.2 | 90.0 | 83.3
  Day 7: number analyzed (Participants) | 39 | 29 | 30
  Day 7 | 76.9 | 79.3 | 76.7
Statistical Analysis 1: Comparison: Pooled Placebo vs AT-527 550 mg (1x550 mg); Day 3; Test type: Superiority; Difference in Percentage of Positivity = 5.00, 80% CI 2-sided [-0.16 to 10.16] — Confidence interval estimated with the Farrington-Manning method
Statistical Analysis 2: Comparison: Pooled Placebo vs AT-527 1100 mg (4x275 mg); Day 3; Test type: Superiority; Difference in Percentage of Positivity = -1.90, 80% CI 2-sided [-9.20 to 5.41] — Confidence interval estimated with the Farrington-Manning method
Statistical Analysis 3: Comparison: Pooled Placebo vs AT-527 550 mg (1x550 mg); Day 5; Test type: Superiority; Difference in Percentage of Positivity = 5.79, 80% CI 2-sided [-4.82 to 16.40] — Confidence interval estimated with the Farrington-Manning method
Statistical Analysis 4: Comparison: Pooled Placebo vs AT-527 1100 mg (4x275 mg); Day 5; Test type: Superiority; Difference in Percentage of Positivity = -0.88, 80% CI 2-sided [-12.40 to 10.65] — Confidence interval estimated with the Farrington-Manning method
Statistical Analysis 5: Comparison: Pooled Placebo vs AT-527 550 mg (1x550 mg); Day 7; Test type: Superiority; Difference in Percentage of Positivity = 2.39, 80% CI 2-sided [-10.64 to 15.42] — Confidence interval estimated with the Farrington-Manning method
Statistical Analysis 6: Comparison: Pooled Placebo vs AT-527 1100 mg (4x275 mg); Day 7; Test type: Superiority; Difference in Percentage of Positivity = -0.26, 80% CI 2-sided [-13.39 to 12.88] — Confidence interval estimated with the Farrington-Manning method

5. Secondary Outcome: Area Under the Curve (AUC) in the Amount of SARS-CoV-2 Virus RNA
Description: AUC is the amount of SARS-CoV-2 virus RNA from baseline to the last sample timepoint and was calculated using the trapezoidal method. RT-PCR was measured from NP swabs.
Time Frame: Baseline, Day 3, Day 5, Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log10 copies/mL*hour
Arm/Group | Pooled Placebo | AT-527 550 mg (1x550 mg) | AT-527 1100 mg (4x275 mg)
Number analyzed (Participants) | 40 | 30 | 30
log10 copies/mL*hour | 651.56 (189.10) | 733.70 (146.63) | 618.62 (194.88)

6. Secondary Outcome: Time to Alleviation or Improvement of COVID-19 Symptoms (21.5 Hours)
Description: COVID-19 symptoms were evaluated using the first 12 items in the COVID-19 Symptom Diary, which included the following 12 items: nasal congestion or runny nose, sore throat, cough, shortness of breath, muscle or body aches, fatigue, headache, chills/sweats, feeling hot or feverish, nausea, vomiting, and diarrhea. The symptoms were scored on the 4-point Likert scale (0=none, 1=mild, 2=moderate, 3=severe).Time to alleviation or improvement is defined as the length of time taken from start of treatment to the point at which all of the following three criteria are met and maintained for a concurrent duration of at least 21.5 hours: "new" symptoms with a score of 0 or 1; "pre- existing and worsened due to COVID-19" symptoms with at least a single category improvement from baseline; "pre-existing and not worsened due to COVID-19" symptoms remaining the same or at least a single category improvement from baseline.
Time Frame: Up to 28 Days
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Pooled Placebo | AT-527 550 mg (1x550 mg) | AT-527 1100 mg (4x275 mg)
Number analyzed (Participants) | 40 | 30 | 30
hours | 43.4 [9.3 to 104.7] | 57.2 [9.0 to 115.8] | 56.4 [2.5 to 96.4]

7. Secondary Outcome: Time to Alleviation or Improvement of COVID-19 Symptoms (43 Hours)
Description: COVID-19 symptoms were evaluated using the first 12 items in the COVID-19 Symptom Diary, which included the following 12 items: nasal congestion or runny nose, sore throat, cough, shortness of breath, muscle or body aches, fatigue, headache, chills/sweats, feeling hot or feverish, nausea, vomiting, and diarrhea. The symptoms were scored on the 4-point Likert scale (0=none, 1=mild, 2=moderate, 3=severe). Time to alleviation or improvement is defined as the length of time taken from start of treatment to the point at which all of the following three criteria are met and maintained for a concurrent duration of at least 43 hours: "new" symptoms with a score of 0 or 1; "pre- existing and worsened due to COVID-19" symptoms with at least a single category improvement from baseline; "pre-existing and not worsened due to COVID-19" symptoms remaining the same or at least a single category improvement from baseline.
Time Frame: Up to 28 Days
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Pooled Placebo | AT-527 550 mg (1x550 mg) | AT-527 1100 mg (4x275 mg)
Number analyzed (Participants) | 40 | 30 | 30
hours | 43.4 [9.3 to 104.7] | 57.2 [9.0 to 141.2] | 58.1 [2.5 to 118.2]

8. Secondary Outcome: Time to Alleviation of COVID-19 Symptoms (21.5 Hours)
Description: COVID-19 symptoms were evaluated using the first 12 items in the COVID-19 Symptom Diary, which included the following 12 items: nasal congestion or runny nose, sore throat, cough, shortness of breath, muscle or body aches, fatigue, headache, chills/sweats, feeling hot or feverish, nausea, vomiting, and diarrhea. The symptoms were scored on the 4-point Likert scale (0=none, 1=mild, 2=moderate, 3=severe). Time to alleviation of COVID-19 symptoms is defined as the length of time taken from start of treatment to the point at which the following criterion is met and maintained for at least 21.5 hours: Score of 0 or 1 on Items 1-12 of the COVID-19 Symptom Diary, regardless of if the symptom is pre-existing or new.
Time Frame: Up to 28 Days
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Pooled Placebo | AT-527 550 mg (1x550 mg) | AT-527 1100 mg (4x275 mg)
Number analyzed (Participants) | 40 | 30 | 30
hours | 43.4 [9.3 to 104.7] | 57.2 [9.0 to 115.8] | 56.4 [8.2 to 96.4]

9. Secondary Outcome: Time to Alleviation of COVID-19 Symptoms (43 Hours)
Description: COVID-19 symptoms were evaluated using the first 12 items in the COVID-19 Symptom Diary, which included the following 12 items: nasal congestion or runny nose, sore throat, cough, shortness of breath, muscle or body aches, fatigue, headache, chills/sweats, feeling hot or feverish, nausea, vomiting, and diarrhea. The symptoms were scored on the 4-point Likert scale (0=none, 1=mild, 2=moderate, 3=severe). Time to alleviation of COVID-19 symptoms is defined as the length of time taken from start of treatment to the point at which the following criterion is met and maintained for at least 43 hours: Score of 0 or 1 on Items 1-12 of the COVID-19 Symptom Diary, regardless of if the symptom is pre-existing or new.
Time Frame: Up to 28 Days
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Pooled Placebo | AT-527 550 mg (1x550 mg) | AT-527 1100 mg (4x275 mg)
Number analyzed (Participants) | 40 | 30 | 30
hours | 43.4 [9.3 to 104.7] | 57.2 [9.0 to 141.2] | 58.1 [8.2 to 118.2]

10. Secondary Outcome: Duration of Fever
Description: Duration of fever was defined as the time from start of treatment to return to an afebrile state (temperature ≤ 37.5°C) maintained for at least 21.5 hours.
Time Frame: Up to 28 Days
Population: The modified ITT infected (mITTi) population was defined as all participants randomized in the study who received any amount of study drug and had at least one positive SARS-CoV-2 RT-PCR test result above or equal to the limit of quantification (LOQ) during the study, with participants grouped according to the treatment assignment at randomization. Only participants who had a fever (temperature > 37.5 degrees Celsius) at baseline are included.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Pooled Placebo | AT-527 550 mg (1x550 mg) | AT-527 1100 mg (4x275 mg)
Number analyzed (Participants) | 2 | 0 | 0
hours | 10.6 [9.6 to 11.7] |  |

11. Secondary Outcome: Percentage of Participants With COVID-19 Related Complications
Description: COVID-19 related complications include death, hospitalization, radiologically confirmed pneumonia, acute respiratory failure, sepsis, coagulopathy, pericarditis, myocarditis, and cardiac failure.
Time Frame: Up to 33 Days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo | AT-527 550 mg (1x550 mg) | AT-527 1100 mg (4x275 mg)
Number analyzed (Participants) | 40 | 30 | 30
percentage of participants | 0 | 3.3 | 3.3

12. Secondary Outcome: Time to Alleviation of an Individual Symptom
Description: The COVID-19 Symptom Diary included the following 14 items: nasal congestion or runny nose, sore throat, cough, shortness of breath, muscle or body aches, fatigue, headache, chills/sweats, feeling hot or feverish, nausea, vomiting, diarrhea, sense of smell over the past 7 days and sense of taste over the past 7 days. The severity of items 1-12 was recorded on a 4-point Likert scale (none=0, mild=1, moderate=2, severe=3). Items 13-14 were recorded on a 3-point Likert scale (same as usual=0, less than usual=1, no sense=2). Time to alleviation of an individual symptom was defined as the time taken from the start of treatment to the point at which the following criterion was met and maintained (for each individual symptom) for at least 21.5 hours: score of 0 or 1 for Items 1-12 of the COVID-19 Symptom Diary; score of 0 for Items 13 and 14 of the COVID-19 Symptom Diary.
Time Frame: Up to 28 Days
Population: The mITTi population was defined as all participants randomized in the study who received any amount of study drug and had at least one positive SARS-CoV-2 RT-PCR test result above or equal to the limit of quantification (LOQ) during the study, with participants grouped according to the treatment assignment at randomization. Only participants with a baseline score of > 1 for Items 1 - 12 or > 0 for Items 13 - 14 of the COVID-19 Symptom Diary were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Pooled Placebo | AT-527 550 mg (1x550 mg) | AT-527 1100 mg (4x275 mg)
Number analyzed (Participants) | 40 | 30 | 30
hours
  Nasal Congestion/Runny Nose: number analyzed (Participants) | 12 | 8 | 10
  Nasal Congestion/Runny Nose | 27.6 [11.3 to 59.9] | 34.2 [15.8 to 82.4] | 32.7 [10.0 to 57.7]
  Sore Throat: number analyzed (Participants) | 5 | 5 | 2
  Sore Throat | 20.5 [14.1 to 22.7] | 24.1 [9.8 to 45.0] | 111.7 [22.1 to 201.4]
  Cough: number analyzed (Participants) | 11 | 6 | 7
  Cough | 22.6 [11.8 to 129.3] | 90.7 [23.7 to 140.4] | 33.9 [20.5 to 119.2]
  Shortness of Breath: number analyzed (Participants) | 3 | 2 | 1
  Shortness of Breath | 23.9 [11.5 to NA] — NA: not estimable due to low number of participants with an event. | 68.9 [68.5 to 69.2] | 11.6 [11.6 to 11.6]
  Aches and Pains: number analyzed (Participants) | 8 | 8 | 4
  Aches and Pains | 33.1 [11.8 to 60.4] | 22.3 [16.3 to 62.2] | 94.4 [48.1 to 177.7]
  Fatigue: number analyzed (Participants) | 15 | 10 | 11
  Fatigue | 47.8 [22.6 to 178.1] | 44.4 [10.5 to 94.5] | 70.6 [22.6 to 106.0]
  Headache: number analyzed (Participants) | 13 | 7 | 11
  Headache | 32.0 [10.1 to 95.8] | 11.7 [9.8 to 93.6] | 34.4 [21.8 to 105.4]
  Chills/Sweats: number analyzed (Participants) | 8 | 3 | 4
  Chills/Sweats | 11.8 [9.8 to 24.1] | 12.0 [9.0 to 35.8] | 25.0 [17.1 to 41.4]
  Feeling Hot or Feverish: number analyzed (Participants) | 6 | 2 | 4
  Feeling Hot or Feverish | 26.5 [11.8 to 35.7] | 48.0 [24.0 to 72.0] | 40.3 [15.9 to 63.4]
  Nausea: number analyzed (Participants) | 2 | 0 | 0
  Nausea | NA [21.1 to NA] — NA: not estimable due to low number of participants with an event. |  |
  Vomiting: number analyzed (Participants) | 2 | 0 | 0
  Vomiting | NA [11.0 to NA] — NA: not estimable due to low number of participants with an event. |  |
  Diarrhea: number analyzed (Participants) | 1 | 0 | 1
  Diarrhea | NA [NA to NA] — NA: not estimable due to low number of participants with an event. |  | 9.8 [9.8 to 9.8]
  Sense of Smell: number analyzed (Participants) | 19 | 14 | 18
  Sense of Smell | 261.5 [164.9 to NA] — NA: not estimable due to low number of participants with an event. | 290.2 [130.7 to NA] — NA: not estimable due to low number of participants with an event. | 213.1 [129.7 to 513.7]
  Sense of Taste: number analyzed (Participants) | 16 | 12 | 17
  Sense of Taste | 221.1 [165.3 to 297.6] | 214.1 [94.1 to NA] — NA: not estimable due to low number of participants with an event. | 178.5 [105.5 to 391.2]

13. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any of the following: any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the medicinal product, any new disease or exacerbation of an existing disease, recurrence of an intermittent medical condition not present at baseline or related to a protocol-mandated intervention.
Time Frame: Up to 33 Days
Population: Safety population consisted of all participants who received any amount of study drug and were grouped according to the treatment that the participants actually received rather than the treatment assigned at randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo | AT-527 550 mg (1x550 mg) | AT-527 1100 mg (4x275 mg)
Number analyzed (Participants) | 40 | 30 | 30
percentage of participants | 27.5 | 20.0 | 33.3

14. Secondary Outcome: Plasma Concentrations of AT-511, AT-551, AT-229 and AT-273 for Participants Treated With 550 mg AT-527
Description: AT-511 is the free base form of AT-527. Its major metabolites are AT-551, AT-229, and AT-273.
Time Frame: Day 1: pre-dose, 1 hour, 3 hours; Day 3: pre-dose; Day 5: pre-dose, 3 hours, 48 hours
Population: The pharmacokinetic-evaluable population consisted of all participants randomized into the study who had at least one post-dose drug concentration measurement at a scheduled visit timepoint.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | AT-527 550 mg (1x550 mg)
Number analyzed (Participants) | 30
nanograms per milliliter (ng/mL)
  AT-511: Day 1, pre-dose | 1.3 (4.5)
  AT-511: Day 1, 1 hour | 1950.5 (2365.0)
  AT-511: Day 1, 3 hours: number analyzed (Participants) | 29
  AT-511: Day 1, 3 hours | 441.4 (645.8)
  AT-511: Day 3, pre-dose: number analyzed (Participants) | 28
  AT-511: Day 3, pre-dose | 254.2 (943.1)
  AT-511: Day 5, pre-dose | 5.6 (21.9)
  AT-511: Day 5, 3 hours | 415.7 (445.5)
  AT-511: Day 5, 48 hours: number analyzed (Participants) | 29
  AT-511: Day 5, 48 hours | 0.5 (0.0)
  AT-551: Day 1, pre-dose | 0.5 (0.0)
  AT-551: Day 1, 1 hour | 347.5 (334.1)
  AT-551: Day 1, 3 hours: number analyzed (Participants) | 29
  AT-551: Day 1, 3 hours | 375.8 (303.9)
  AT-551: Day 3, pre-dose: number analyzed (Participants) | 28
  AT-551: Day 3, pre-dose | 56.9 (100.1)
  AT-551: Day 5, pre-dose | 26.6 (22.7)
  AT-551: Day 5, 3 hours | 323.8 (168.3)
  AT-551: Day 5, 48 hours: number analyzed (Participants) | 29
  AT-551: Day 5, 48 hours | 1.7 (1.4)
  AT-229: Day 1, pre-dose | 0.5 (0.0)
  AT-229: Day 1, 1 hour | 268.5 (318.5)
  AT-229: Day 1, 3 hours: number analyzed (Participants) | 29
  AT-229: Day 1, 3 hours | 427.4 (275.8)
  AT-229: Day 3, pre-dose: number analyzed (Participants) | 28
  AT-229: Day 3, pre-dose | 290.3 (152.3)
  AT-229: Day 5, pre-dose | 295.4 (145.0)
  AT-229: Day 5, 3 hours | 773.9 (340.8)
  AT-229: Day 5, 48 hours: number analyzed (Participants) | 29
  AT-229: Day 5, 48 hours | 89.2 (87.8)
  AT-273: Day 1, pre-dose | 0.5 (0.0)
  AT-273: Day 1, 1 hour | 26.5 (29.0)
  AT-273: Day 1, 3 hours: number analyzed (Participants) | 29
  AT-273: Day 1, 3 hours | 132.2 (66.7)
  AT-273: Day 3, pre-dose: number analyzed (Participants) | 28
  AT-273: Day 3, pre-dose | 135.9 (47.6)
  AT-273: Day 5, pre-dose | 138.1 (53.0)
  AT-273: Day 5, 3 hours | 236.9 (79.9)
  AT-273: Day 5, 48 hours: number analyzed (Participants) | 29
  AT-273: Day 5, 48 hours | 40.9 (22.7)

15. Secondary Outcome: Plasma Concentrations of AT-511, AT-551, AT-229 and AT-273 for Participants Treated With 1100 mg AT-527
Description: AT-511 is the free base form of AT-527. Its major metabolites are AT-551, AT-229, and AT-273.
Time Frame: Day 1: pre-dose, 1 hour, 4 hours; Day 3: pre-dose; Day 5: pre-dose, 1 hour, 4 hours, 48 hours
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | AT-527 1100 mg (4x275 mg)
Number analyzed (Participants) | 30
nanograms per milliliter (ng/mL)
  AT-511: Day 1, pre-dose: number analyzed (Participants) | 29
  AT-511: Day 1, pre-dose | 0.5 (0.0)
  AT-511: Day 1, 1 hour: number analyzed (Participants) | 29
  AT-511: Day 1, 1 hour | 3575.0 (2883.6)
  AT-511: Day 1, 4 hours | 852.4 (1513.2)
  AT-511: Day 3, pre-dose: number analyzed (Participants) | 24
  AT-511: Day 3, pre-dose | 9.6 (15.9)
  AT-511: Day 5, pre-dose: number analyzed (Participants) | 26
  AT-511: Day 5, pre-dose | 316.7 (1544.7)
  AT-511: Day 5, 1 hour: number analyzed (Participants) | 25
  AT-511: Day 5, 1 hour | 3568.9 (3352.1)
  AT-511: Day 5, 4 hours: number analyzed (Participants) | 23
  AT-511: Day 5, 4 hours | 1323.3 (2883.5)
  AT-511: Day 5, 48 hours: number analyzed (Participants) | 24
  AT-511: Day 5, 48 hours | 0.6 (0.6)
  AT-551: Day 1, pre-dose: number analyzed (Participants) | 29
  AT-551: Day 1, pre-dose | 0.5 (0.0)
  AT-551: Day 1, 1 hour: number analyzed (Participants) | 29
  AT-551: Day 1, 1 hour | 592.2 (576.9)
  AT-551: Day 1, 4 hours | 640.4 (446.3)
  AT-551: Day 3, pre-dose: number analyzed (Participants) | 25
  AT-551: Day 3, pre-dose | 84.0 (72.1)
  AT-551: Day 5, pre-dose: number analyzed (Participants) | 26
  AT-551: Day 5, pre-dose | 71.3 (61.6)
  AT-551: Day 5, 1 hour: number analyzed (Participants) | 25
  AT-551: Day 5, 1 hour | 302.8 (222.1)
  AT-551: Day 5, 4 hours: number analyzed (Participants) | 23
  AT-551: Day 5, 4 hours | 342.1 (254.9)
  AT-551: Day 5, 48 hours: number analyzed (Participants) | 24
  AT-551: Day 5, 48 hours | 4.4 (4.8)
  AT-229: Day 1, pre-dose: number analyzed (Participants) | 29
  AT-229: Day 1, pre-dose | 0.5 (0.0)
  AT-229: Day 1, 1 hour: number analyzed (Participants) | 29
  AT-229: Day 1, 1 hour | 371.9 (460.3)
  AT-229: Day 1, 4 hours | 865.4 (494.2)
  AT-229: Day 3, pre-dose: number analyzed (Participants) | 25
  AT-229: Day 3, pre-dose | 682.8 (351.7)
  AT-229: Day 5, pre-dose: number analyzed (Participants) | 26
  AT-229: Day 5, pre-dose | 797.8 (459.9)
  AT-229: Day 5, 1 hour: number analyzed (Participants) | 25
  AT-229: Day 5, 1 hour | 990.9 (505.3)
  AT-229: Day 5, 4 hours: number analyzed (Participants) | 23
  AT-229: Day 5, 4 hours | 1357.2 (825.3)
  AT-229: Day 5, 48 hours: number analyzed (Participants) | 24
  AT-229: Day 5, 48 hours | 279.4 (285.3)
  AT-273: Day 1, pre-dose: number analyzed (Participants) | 29
  AT-273: Day 1, pre-dose | 0.5 (0.0)
  AT-273: Day 1, 1 hour: number analyzed (Participants) | 29
  AT-273: Day 1, 1 hour | 35.7 (47.4)
  AT-273: Day 1, 4 hours | 231.8 (111.4)
  AT-273: Day 3, pre-dose: number analyzed (Participants) | 25
  AT-273: Day 3, pre-dose | 245.6 (122.8)
  AT-273: Day 5, pre-dose: number analyzed (Participants) | 26
  AT-273: Day 5, pre-dose | 263.6 (107.3)
  AT-273: Day 5, 1 hour: number analyzed (Participants) | 25
  AT-273: Day 5, 1 hour | 252.1 (97.4)
  AT-273: Day 5, 4 hours: number analyzed (Participants) | 23
  AT-273: Day 5, 4 hours | 310.6 (107.5)
  AT-273: Day 5, 48 hours: number analyzed (Participants) | 24
  AT-273: Day 5, 48 hours | 84.4 (45.5)

16. Primary Outcome: Change From Baseline in the Amount of Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Virus RNA for AT-527 1100 mg and Pooled Placebo
Description: SARS-CoV-2 virus RNA was measured by reverse-transcription polymerase chain reaction (RT-PCR) from NP swabs. The change from baseline was estimated from an ANCOVA model with baseline viral load as a covariate. Reported here is the adjusted mean change from baseline. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Day 3, Day 5, Day 7
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Pooled Placebo | AT-527 1100 mg (4x275 mg)
Number analyzed (Participants) | 40 | 30
log10 copies/mL
  Day 3: number analyzed (Participants) | 40 | 29
  Day 3 | -1.08 (0.190) | -1.18 (0.223)
  Day 5: number analyzed (Participants) | 38 | 30
  Day 5 | -2.21 (0.205) | -2.31 (0.231)
  Day 7: number analyzed (Participants) | 39 | 30
  Day 7 | -2.70 (0.207) | -2.78 (0.236)
Statistical Analysis 1: Comparison: Pooled Placebo vs AT-527 1100 mg (4x275 mg); Day 3; Test type: Superiority; p = 0.7351, ANCOVA; Difference in Adjusted Means = -0.10, 80% CI 2-sided [-0.48 to 0.28], Standard Error of Mean 0.294 — A difference in adjusted means of <0 favors RO7496998 (AT-527)
Statistical Analysis 2: Comparison: Pooled Placebo vs AT-527 1100 mg (4x275 mg); Day 5; Test type: Superiority; p = 0.7524, ANCOVA; Difference in Adjusted Means = -0.10, 80% CI 2-sided [-0.50 to 0.30], Standard Error of Mean 0.310 — A difference in adjusted means of <0 favors RO7496998 (AT-527)
Statistical Analysis 3: Comparison: Pooled Placebo vs AT-527 1100 mg (4x275 mg); Day 7; Test type: Superiority; p = 0.8083, ANCOVA; Difference in Adjusted Means = -0.08, 80% CI 2-sided [-0.48 to 0.33], Standard Error of Mean 0.314 — A difference in adjusted means of <0 favors RO7496998 (AT-527)

ADVERSE EVENTS:
Time Frame: Up to 33 days
Description: Safety Population consisted of all participants who received any amount of study drug and were grouped according to the treatment that the participants actually received rather than the treatment assigned at randomization.
Arm/Group | Pooled Placebo | AT-527 550 mg (1x550 mg) | AT-527 1100 mg (4x275 mg)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/40 | 1/30 | 1/30
Other Adverse Events (participants affected / at risk) | 1/40 | 1/30 | 5/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled Placebo (N=40) | AT-527 550 mg (1x550 mg) (N=30) | AT-527 1100 mg (4x275 mg) (N=30)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled Placebo (N=40) | AT-527 550 mg (1x550 mg) (N=30) | AT-527 1100 mg (4x275 mg) (N=30)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT04709835/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT04709835/SAP_001.pdf